CLINICAL TRIAL: NCT05251389
Title: Conversion of Unresponsiveness to Immunotherapy by Fecal Microbiota Transplantation in Patients With Metastatic Melanoma: a Randomized Phase Ib/IIa Trial
Brief Title: FMT to Convert Response to Immunotherapy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N21FMT
Record Dates: First submitted 2021-12-20; First posted 2022-02-22 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Melanoma Stage III; Melanoma Stage IV
MeSH Terms: conditions — Melanoma | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: a randomized double-blind intervention trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: FMT from an ICI non-responding donor (Experimental): Patients will receive FMT from an ICI non-responding donor (defined as ≥20% increase according to RECIST 1.1 criteria within the past 3 months). Patients will continue their anti-PD-1 treatment.
  Interventions: Other: Fecal microbiota transplantation
- B: FMT from an ICI responding donor (Experimental): Patients will receive FMT from an ICI responding donor (defined as ≥30% decrease or disappearance of all lesions according to RECIST 1.1 criteria within the past 24 months). Patients will continue their anti-PD-1 treatment.
  Interventions: Other: Fecal microbiota transplantation

INTERVENTIONS:
Other: Fecal microbiota transplantation — Fecal microbiota transplantation of an ICI responding or Fecal microbiota transplantation from an ICI non-responding donor, in combination with ICI.

SUMMARY:
In this study the aim is to investigate whether transfer of the microbiota of either responder or non-responder patients via fecal microbiotica transplantation (FMT) can convert the response to immunotherapy in immune checkpoint inhibitors (ICI) refractory metastatic melanoma patients.

This is a randomized double-blind intervention phase Ib/IIa trial in ICI refractory metastatic melanoma patients receiving either FMT of an ICI responding or FMT from an ICI non-responding donor, in combination with ICI.

Following randomization, patients will receive vancomycin 250 mg, four times daily for 4 days (day -5 up until day -2), and undergo bowel clearance on day -1 (in total 1L MoviPrep). The FMT, either derived from donor group R (who showed a good response on anti-PD-1 therapy) or donor group NR (who showed progression on anti-PD-1 therapy), will be performed by a gastroenterologist using esophagogastroduodenoscopy. A total amount of 198mL (containing a total of 60 gram feces) will be used for transplantation. Anti-PD-1 treatment will be continued according to the patient's regular treatment schedule. Evaluation of safety and response to treatment will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be 18 years or older
* Patients have pathologically confirmed advanced stage cutaneous melanoma (stage III or IV) requiring systemic treatment with anti-PD-1

  * In case of stage IV disease, only patients with M1a or M1b disease are eligible.
* Patients have confirmed disease progression (≥20% increase according to RECIST1.1) on two consecutive scans with a four week interval while on anti-PD-1 treatment, of which the second scan has to be performed within 3 weeks prior to signing informed consent.
* Patients must have measurable disease per RECIST 1.1 criteria
* Patients have an ECOG performance status of 0-1 (appendix D)
* Patients have a life expectancy of >3 months
* Patients have adequate organ function as determined by standard-of-care pre-checkpoint inhibitor infusion lab (including serum ALAT/ASAT less than three times the upper limit of normal (ULN); serum creatinine clearance 50ml/min or higher; total bilirubin less than or equal to 20 micromol/L, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 50 micromol/L)
* Patients have an LDH level of ≤1 times ULN
* Patients of both genders must be willing to use a highly effective method of birth control during treatment
* Patients must be able to understand and sign the Informed Consent document

Exclusion Criteria:

* Patients with acral, uveal or mucosal melanoma, or patients with an unknown primary
* Patients who have received treatment for their melanoma other than anti-PD-1 treatment.
* Stage IV patients with M1c or M1d disease.
* Patients with autoimmune diseases: patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's disease, are excluded from this study (except Hashimoto thyroiditis, vitiligo, history of psoriasis, but no active disease)
* Patients with any grade 3 or 4 immune-related adverse events still requiring active immunosuppressive medication, apart from endocrinopathies that are stable under hormone replacement therapy. Patients who had developed grade 3-4 immune related toxicity, which has reverted to grade I with immunosuppressive drugs and who are off immunosuppression at least two weeks prior to enrollment are eligible
* Patients with brain or LM metastasis.
* Patients with an elevated LDH level
* Patients that have undergone major gastric/esophageal/bowel surgery (like Wipple, subtotal colectomy)
* Severe food allergy (e.g. nuts, shellfish)
* Patients with a swallowing disorder or expected bowel passage problems (ileus, fistulas, perforation)
* Severe dysphagia with incapability of swallowing 2 liters of bowel lavage
* Patients with a life expectancy of less than three months
* Patients with severe cardiac or pulmonary comorbidities (per judgement of the investigator)
* Women who are pregnant or breastfeeding
* Patients with any active systemic infections, coagulation disorders or other active major medical illnesses
* Patients with other malignancies, except adequately treated and a cancer-related life-expectancy of more than 5 years
* Patients who received treatment with antibiotics in the three months prior to study enrolment, or patients we are expected to receive systemic antibiotics during the course of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Efficacy, defined as clinical benefit (stable disease (SD), partial response (PR), complete response (CR) | At 12 weeks after FMT

SECONDARY OUTCOMES:
Safety, measured as the occurrence of toxicity of grade 3 or higher | At screening, and 2 weeks, 6 weeks, 12 weeks and 16 weeks after FMT
Progression free survival (PFS) | Up to one year post-FMT
  PFS will be calculated from the date of registration to the date of progression or death, whichever occurs first, censoring patients without progression and who are still alive at last follow-up
The change in gut microbiome following FMT and the duration and stability over time | At screening, and 2 weeks, 6 weeks, 12 weeks and 16 weeks after FMT
  To assess the fecal microbiome (which includes bacteria, archaea, viruses, parasites and fungi), nucleotides will be isolated for next generation sequencing and molecular methodologies (e.g. PCR, qPCR). Initially, whole genomic DNA (metagenomics) and the ITS2 region or the rRNA gene will be will be sequenced, giving insights in the overall microbiota's structural and functional features and in the structural features of the fungal microbiota, respectively, which both will be associated to clinical variables.
The change in metabolome following FMT and the duration and stability over time | At screening, and 2 weeks, 6 weeks, 12 weeks and 16 weeks after FMT
  To assess the metabolome in feces (which includes amino acids, short lipids, sugars and nucleotides), samples will be processed and analyzed by Liquid Chromatography Tandem Mass Spectrometry (LC-MS/MS) or Nuclear magnetic resonance (NMR). The identified metabolic profile will be associated with the microbiome data and clinical variables.
The immune changes; changes in cell populations (absolute, relative, phenotypical), in chemokine/cytokine levels and in the tumor-microenvironment | At screening, and 2 weeks, 6 weeks, 12 weeks and 16 weeks after FMT
  Tumor biopsies and blood samples will be analyzed to investigator the local and systemic immune changes: changes in cell populations (absolute, relative, phenotypical), in chemokine/cytokine levels and in the tumor-microenvironment (TME). If possible, results will be linked to response.

CONTACTS AND LOCATIONS:
Overall Officials: John Haanen, Prof, Principal Investigator — Medical Oncologist
Locations (1):
- Antoni van Leeuwenhoek, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Borgers JSW, Burgers FH, Terveer EM, van Leerdam ME, Korse CM, Kessels R, Flohil CC, Blank CU, Schumacher TN, van Dijk M, Henderickx JGE, Keller JJ, Verspaget HW, Kuijper EJ, Haanen JBAG. Conversion of unresponsiveness to immune checkpoint inhibition by fecal microbiota transplantation in patients with metastatic melanoma: study protocol for a randomized phase Ib/IIa trial. BMC Cancer. 2022 Dec 30;22(1):1366. doi: 10.1186/s12885-022-10457-y. PMID 36585700